CLINICAL TRIAL: NCT05876650
Title: Compariso of Pilates Exercises and Yoga on Rounded Shoulders
Brief Title: Pilates Exercises v/s Yoga on Rounded Shoulders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIPHAH/FR&AHS/Letter-014121
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Weakness, Muscle; Muscle Tightness; Range of Motion; Pain; Heart Rate; SpO2; Sleep Quality
MeSH Terms: conditions — Muscle Weakness; Pain; Sleep Initiation and Maintenance Disorders | interventions — Exercise Movement Techniques; Yoga

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise Group (Experimental): 6 Pilates exercises that are Swan, Swimming, Prone press up, Dart, Arm arch and Scarecow.
  Interventions: Other: Pilates exercises
- Yoga Group (Experimental): 6 Yoga poses: Warrior pose 1, Triangle pose, Child pose, Cow face pose, Bound angle pose, half bow pose.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Pilates exercises — Pilates exercises starts with warm up, followed by 6 main exercises that are Swan, Swimming, Prone press up, Dart, Arm arch and Scarecow. The session will end with the cool down exercises. Each exercise will be repeated 10 times for 5 sets. Patients will be treated 3 times per week for 4 consecutive weeks.
  Arms: Pilates exercise Group
Other: Yoga — Yoga will start with warm up followed by 6 yoga poses which are Warrior pose 1, Triangle pose, Child pose, Cow face pose, Bound angle pose, half bow poseThe session will end with a cool down pose. Each yoga pose will be held for 8-10 breathes Patients will be treated 3 times per week for 4 consecutive weeks.
  Arms: Yoga Group

SUMMARY:
To Compare the effects of Pilates exercises an yoga on rounded shoulders

DETAILED DESCRIPTION:
Pilates exercises and Yoga are two effective treatments for correcting RSP. In Pilates each exercise is conducted in more than one times usually three to five hence exposing the body to different and new muscular and kinesthetic challenges. On the other hand Yoga is a process in which the joints and muscles operate together in a systematic and automatic manner where each pose is sustained for a period of time. Several literatures support the belief that Pilates exercises and Yoga are effective treatments for RSP correction, as well as improving sleep quality, heart rate and SpO2 First, The participants will be divided into two groups, for Pilates exercises and Yoga. Honor wristbands will be distributed and Exercises will be demonstrated to each group. Explanation of using Honor band will be given. Measurements will be taken before the intervention including cervical ROM. shoulder ROM at baseline, 2nd week and 4th week. while heart rate, SpO2 immediately after the session. Sleep quality prior the intervention, 2nd and 4th week. Patients will do the exercises 3 times per week for 4 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rounded shoulders who achieve more than 2.5 cm in table top test.

Exclusion Criteria:

* Patients with a positive history of trauma, fracture or surgery of the cervical spine or shoulder.
* Neck pain with radiation to the arm and upper extremity.
* Diagnosed cases of torticollis and scoliosis.
* Patient with any serious underlying pathology that influence the mobility of upper limb
* History of osteoporosis, any heart disease

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Rigid transparent plastic protractor | 2nd week and 4th week
  changes from baseline measurement of the distance between the posterior border of the acromion and the wall or a table

SECONDARY OUTCOMES:
Neck diability Index | 4th week
  Changes from baseline The neck disability index is a ten-item self-reported questionnaire that assesses pain and associated disability, with a total max score of 50 points. he NDI consists of 10 domains-pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleep, and recreation-designed to assess the level of disability in patients with neck pain.
Goniometer | 2nd week and 4th week
  Changes from baseline Measurements of cervical flexion, extension, lateral flexion, and rotation, Shoulder flexion, extension, abduction, adduction, internal and external rotation were found to be reliable with universal goniometer
The Shoulder Pain and Disability Index | 4th week
  Change from baseline SPADI is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The SPADI includes two domains: a five-item pain subscale and an eight-item disability subscale. he maximum score is 130
Honor Band 5 Smart Wristband Fitness Tracker | 2nd week and 4th week
  Changes from baseline With optimized optical hardware and software algorithms, HONOR Band 5 precisely measure, HR , SpO2 both immediately after exercise and monitors sleep throughout the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PHD*, Principal Investigator — Riphah College of Rehabilitation and Allied Health Sciences, Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No